CLINICAL TRIAL: NCT07226648
Title: Ultrasonic Neuromodulation of Cingulate Cortex for Fibromyalgia: A Blinded Randomized Sham-Controlled Trial
Brief Title: Ultrasonic Neuromodulation of Cingulate Cortex for Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SPIRE Therapeutics Inc. (Industry)
Collaborators: University of Utah Data Coordinating Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPIRE1002025
Record Dates: First submitted 2025-11-07; First posted 2025-11-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Focused Ultrasound (Active Comparator)
  Interventions: Device: Focused Ultrasound
- Sham Ultrasound (Sham Comparator)
  Interventions: Device: Focused Ultrasound

INTERVENTIONS:
Device: Focused Ultrasound — DIADEM device

SUMMARY:
The goal of this clinical trial is to evaluate a new noninvasive brain stimulation intervention for fibromyalgia and to determine its effectiveness in reducing pain. Participants will receive four treatments over the course of one month and will complete surveys at multiple time points throughout the 16-week study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent.
2. Age ≥ 22 years.
3. Meets 2016 American College of Rheumatology criteria for fibromyalgia:

   1. Generalized pain, defined as pain in at least 4 of 5 regions, is present, AND
   2. Widespread pain index (WPI) ≥ 7 and symptom severity scale score (SSS) ≥ 5, or WPI of 4-6 and SSS score ≥ 9, AND
   3. Symptoms have been present at a similar level for at least 3 months, AND
   4. A diagnosis of fibromyalgia is valid irrespective of other diagnoses. A diagnosis of fibromyalgia does not exclude the presence of other clinically important illnesses.
4. Failure of at least two evidence-based medications (i.e., pregabalin, duloxetine, milnacipran) for the treatment of fibromyalgia.
5. Failure of one or more attempts at physical or Cognitive Behavioral Therapy (CBT) including:

   1. Aerobic exercise like walking, cycling, and swimming,
   2. Water therapy/hydrotherapy with warm water exercises,
   3. Tai Chi involving slow, controlled movements,
   4. Yoga,
   5. Resistance training,
   6. Bodyweight exercises,
   7. Pilates,
   8. Myofascial release therapy applying gentle pressure on trigger points,
   9. Massage therapy,
   10. Trigger point therapy targeting specific pain points,
   11. Joint mobilization,
   12. Postural retraining to correct body alignment,
   13. Balance and coordination exercises,
   14. Feldenkrais method for movement awareness,
   15. Alexander technique to enhance posture and movement efficiency,
   16. Transcutaneous Electrical Nerve Stimulation (TENS) for pain relief,
   17. Heat therapy using hot packs, infrared, or paraffin wax,
   18. Cold therapy with ice packs or cryotherapy,
   19. Ultrasound therapy for deep tissue relaxation,
   20. Biofeedback to control muscle tension and pain response,
   21. Gentle static stretching for prolonged duration,
   22. Active dynamic stretching for full range of motion,
   23. Proprioceptive Neuromuscular Facilitation (PNF) stretching,
   24. Hydrotherapy pool exercises,
   25. Ai Chi (water-based Tai Chi),
   26. Underwater treadmill therapy, aa) Graded motor imagery (GMI), bb) Mirror therapy to retrain brain-body connections, cc) Mindfulness-based stress reduction (MBSR) combining meditation and movement, dd) Balance exercises to improve stability, ee)Gaze stabilization techniques for dizziness and disorientation, ff) CBT.
6. Pain score of ≥ 4 on Numerical Rating Scale (NRS-11) at Screening visit.
7. Pain score of ≥ 4 on NRS-11 at Baseline visit averaged over 3 consecutive calendar days.
8. Stated willingness and ability to comply with all study procedures.
9. Has remained on the same psychiatric treatment regimen (e.g., medication, psychotherapy) for at least one (1) month prior to screening, and has stated willingness to remain on the same regimen for the duration of the study unless a change in treatment is recommended or agreed upon by the site investigator.
10. For participants who could potentially become pregnant: negative urine pregnancy test at screening; agreement to use a highly effective method of contraception (≤ 1% pregnancy rate) including tubal ligation, vasectomized partner, IUD or IUS (intrauterine device or system), or long-acting contraceptives (LARC).

Exclusion Criteria:

1. Any previous diagnosis of bipolar disorder or schizophrenia-spectrum disorder during the participant's lifetime, according to Diagnostic and Statistical Manual of Mental Disorders, version 5 (DSM-5-TR) criteria.
2. New or existing diagnosis of moderate or severe alcohol or other substance use disorder in the past 6 months, according to DSM-5-TR criteria.
3. New or existing diagnosis of obsessive-compulsive disorder and/or posttraumatic stress disorder in the past 30 days, according to DSM-5-TR criteria, and which is unstable in the clinical judgment of the investigator.
4. New or existing primary diagnosis of anorexia nervosa, bulimia nervosa, or binge eating disorder in the past 3 months, according to DSM-5-TR criteria.
5. Clinically significant neurodevelopmental, neurocognitive, or personality disorder, according to DSM-5-TR criteria.
6. Moderate-High Risk of Suicide, according to the Columbia-Suicide Severity Rating Scale (C-SSRS) Screen Version - Recent (i.e., answers YES to Question 3 and NO to Question 6 (Moderate Risk), or YES to Question 4, 5, or 6 (High Risk)), or in the clinical judgement of the site investigator.
7. Lifetime history of a serious suicide attempt in the medical opinion of the site investigator.
8. Changes in treatment for pain in the past 2 months.
9. Treatment with electroconvulsive therapy, transcranial magnetic stimulation, ketamine, or esketamine in the past 30 days.
10. Currently diagnosed progressive neurological disease such as multiple sclerosis, chronic inflammatory demyelinating polyneuropathy, rapid progressive arachnoiditis, brain or spinal cord tumor, or severe/critical spinal stenosis (stenosis).
11. Cancer-related pain.
12. Diagnosis of malignancy other than basal cell carcinoma, or carcinoma in situ of the cervix within the past five years, to include life expectancy less than one year due to advanced malignancy.
13. Autoimmune-related pain.
14. Inadequately managed general medical condition, in the opinion of the site investigator.
15. Lifetime history of cerebral small vessel disease.
16. Lifetime history of intracranial hemorrhage.
17. Pregnant or breast feeding.
18. Implanted medical device in the head or neck.
19. MRI contraindication or intolerance.
20. Previously enrolled in a DIADEM clinical trial. Note: a patient who screen fails is able to be rescreened at most one time.
21. Has a history of any medical or psychiatric disorder, disease, condition, injury, symptoms, or circumstance that, in the opinion of the site investigator, may (1) reduce the participant's ability to fulfill the study requirements as per protocol; (2) adversely impact the integrity of the data or the validity of the study results; or (3) pose an increased risk to the participant during study participation.
22. Participants with braids, dreadlocks, or other hairstyles that prevent access to the side of the head and who are unwilling to temporarily adjust their hairstyle to allow such access.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale - 11 (NRS-11) pain score | 28 days following initial treatment
  The NRS-11 is a scale from 0-10 with higher values representing higher levels of pain.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire Revised (FIQR) | 28 days following initial treatment
  The FIQR is a scale ranging from 0 to 100 that evaluates function, overall impact, and symptoms of fibromyalgia over the past 7 days. Higher scores represent more severe impact to the patient.
Numerical Rating Scale - 11 (NRS-11) pain score response rate | 28 days following initial treatment
  ≥ 30% reduction from baseline in NRS-11 score (the NRS-11 is a scale from 0-10 with higher values representing higher levels of pain).
Patient-Reported Outcomes Measurement Information System (PROMIS-29) - Pain Interference Subscale | 28 days following initial treatment
  The PROMIS-29 is a 29 question survey assessing physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, and pain intensity. The Pain Interference Subscale is scored on a 5 point scale and asks how much pain interfered with different activities (1 - Not at all; 2 - A little bit; 3 - Somewhat; 4 - Quite a bit; 5 - Very much). Scores are calculated as T-scores with a mean of 50 and a standard deviation of 10. Higher scores represent more pain interference.
Numerical Rating Scale - 11 (NRS-11) pain score response rate | 7 days following initial treatment
  ≥ 30% reduction from baseline in NRS-11 score (the NRS-11 is a scale from 0-10 with higher values representing higher levels of pain).
Patient Global Impression of Improvement (PGI-I) | 28 days following initial treatment
  The PGI-I is a scale from 1-7 indicating how the patient has felt overall since beginning treatment. 1 - Very Much Improved; 2 - Much Improved; 3 - Minimally Improved; 4 - No Change; 5 - Minimally Worse; 6 - Much Worse; 7 - Very Much Worse.
Patient Health Questionnaire-9 (PHQ-9) | 28 days following initial treatment
  The PHQ-9 is a 9-question survey asking "Over the last 2 weeks, how often have you been bothered by any of the following problems?" Each question is scored as:
  0: Not at all;
  1. Several days;
  2. More than half the days;
  3. Nearly every day. The 9 scores are added together, and the total score ranges from 0 to 27, with higher numbers representing more bothersome problems.
Numerical Rating Scale - 11 (NRS-11) pain score | 16 weeks following initial treatment
  The NRS-11 is a scale from 0-10 with higher values representing higher levels of pain.

OTHER OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS-29) - all subscales, excluding Pain Interference | 28 days following initial treatment
  The PROMIS-29 is a 29 question survey assessing physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, and pain intensity. Scores for subscales are calculated as T-scores with a mean of 50 and a standard deviation of 10. Higher scores represent worse health than average for anxiety, depression, fatigue, sleep disturbance, and pain interference. Higher scores represent better health than average for physical function and ability to participate in social roles and activities.
Brief Pain Inventory (BPI) - short form | 28 days following initial treatment
  The BPI includes questions on a scale from 0-10 with higher values representing higher levels of pain or higher levels of pain interference.
Fibromyalgia Impact Questionnaire Revised (FIQR) | 16 weeks following initial treatment
  The FIQR is a scale ranging from 0 to 100 that evaluates function, overall impact, and symptoms of fibromyalgia over the past 7 days. Higher scores represent more severe impact to the patient.
Patient-Reported Outcomes Measurement Information System (PROMIS-29) - all subscales | 16 weeks following initial treatment
  The PROMIS-29 is a 29 question survey assessing physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, and pain intensity. Scores for subscales are calculated as T-scores with a mean of 50 and a standard deviation of 10. Higher scores represent worse health than average for anxiety, depression, fatigue, sleep disturbance, and pain interference. Higher scores represent better health than average for physical function and ability to participate in social roles and activities.
Patient Health Questionnaire-9 (PHQ-9) | 16 weeks following initial treatment
  The PHQ-9 is a 9-question survey asking "Over the last 2 weeks, how often have you been bothered by any of the following problems?" Each question is scored as:
  0: Not at all;
  1. Several days;
  2. More than half the days;
  3. Nearly every day. The 9 scores are added together, and the total score ranges from 0 to 27, with higher numbers representing more bothersome problems.
Patient Global Impression of Improvement (PGI-I) | 16 weeks following initial treatment
  The PGI-I is a scale from 1-7 indicating how the patient has felt overall since beginning treatment. 1 - Very Much Improved; 2 - Much Improved; 3 - Minimally Improved; 4 - No Change; 5 - Minimally Worse; 6 - Much Worse; 7 - Very Much Worse.
Brief Pain Inventory (BPI) - short form | 16 weeks following initial treatment
  The BPI includes questions on a scale from 0-10 with higher values representing higher levels of pain or higher levels of pain interference.
Adverse Events (AEs) | Through 28 days following initial treatment
Serious Adverse Events (SAEs) | Through 16 weeks following initial treatment
Columbia Suicide Severity Rating Scale (C-SSRS) | 28 days following initial treatment
  The C-SSRS is a semi-structured interview to assess suicidal ideation and behavior. Based on responses, participants are categorized as Low Risk, Moderate Risk, or High Risk. An increase in risk level will be evaluated.
Montreal Cognitive Assessment (MoCA) | 28 days following initial treatment
  The MoCA is a neuropsychological screening test with scores ranging from 0-30 with lower scores suggesting higher cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Akiko Okifuji, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Riis TS, Losser AJ, Kassavetis P, Moretti P, Kubanek J. Noninvasive modulation of essential tremor with focused ultrasonic waves. J Neural Eng. 2024 Feb 27;21(1). doi: 10.1088/1741-2552/ad27ef. PMID 38335553
- [Background] Riis TS, Feldman DA, Losser AJ, Okifuji A, Kubanek J. Noninvasive targeted modulation of pain circuits with focused ultrasonic waves. Pain. 2024 Dec 1;165(12):2829-2839. doi: 10.1097/j.pain.0000000000003322. Epub 2024 Jul 30. PMID 39073370
- [Background] Riis TS, Feldman DA, Kwon SS, Vonesh LC, Koppelmans V, Brown JR, Solzbacher D, Kubanek J, Mickey BJ. Noninvasive Modulation of the Subcallosal Cingulate and Depression With Focused Ultrasonic Waves. Biol Psychiatry. 2025 Apr 15;97(8):825-834. doi: 10.1016/j.biopsych.2024.09.029. Epub 2024 Oct 11. PMID 39396736